CLINICAL TRIAL: NCT04159064
Title: Impact of Cardiac Surgery With a Minimal Invasive Extracorporeal Circuit οn Coagulation: Data From Point of Care Testing With Thromboelastometry and Impedance Aggregometry
Brief Title: Impact of Cardiac Surgery With a Minimal Invasive Extracorporeal Circuit οn Coagulation: Data From Point of Care Devices
Status: Completed | Type: Observational
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Eleni Argyriadou, Associate Professor, AHEPA University Hospital
Other Study IDs: 49886/8.11.2018
Record Dates: First submitted 2019-10-21; First posted 2019-11-12 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Extracorporeal Circulation; Complications; Coagulation Disorder; Extracorporeal Circulation of Blood; Thrombocytopenia
Keywords: extracorporeal circulation; coagulation disorder; Extracorporeal Circulation of Blood; Thrombocytopenia
MeSH Terms: conditions — Hemostatic Disorders; Thrombocytopenia | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Minimal Invasive Extracorporeal Circulation(MIECC): Monitoring coagulation using thromboelastometry and platelet function using impedance aggregometry. Samples at the following phases:
  Time 0: Baseline, upon arrival at the operation room (samples for thromboelastometry and impedance aggregometry), Time 2: after aortic cross clamp off (only sample for thromboelastometry), Time 2': 20 minutes post protamine administration (only sample for impedance aggregometry ).
  Interventions: Diagnostic Test: Thromboelastometry, Impedance Aggregometry

INTERVENTIONS:
Diagnostic Test: Thromboelastometry, Impedance Aggregometry — Study of coagulation changes after cardiac surgery on CPB using Minimal Extracorporeal Circulation
  Other Names: Rotational ThromboElastoMetry (ROTEM), ROTEM Platelet

SUMMARY:
This study includes patients undergoing elective cardiac surgery on MiECC. Coagulation status is assessed with ROTEM (TEM International GmbH, Munich, Germany) and Platelet function with impedance aggregometry using the ROTEM-Platelet (TEM International GmbH, Munich, Germany).

DETAILED DESCRIPTION:
Last update: 24th October 2019, Thessaloniki, Greece

Study protocol Objective Abnormal platelet function remains one of the main causes of severe bleeding during cardiac surgery, especially in the era of widespread evolution in antiplatelet therapy as standard of care in cardiac surgery patients. Additionally, conventional cardiopulmonary bypass is identified as a significant attributor to pathophysiologic derangement in coagulation and platelet dysfunction, induced by prolonged contact of blood with foreign surfaces, severe haemodilution, hypothermia and systemic inflammatory response. Minimally invasive extracorporeal circulation (MiECC) reflects the technological progress in cardiopulmonary circuits and offers improved perfusion conditions. The multiple electrode platelet aggregometry analysis can be a useful point-of-care diagnostic tool, assessing platelet receptors inhibition and aggregation, thus providing real-time information perioperatively. Our objective is to investigate the potential protective effect of MiECC on coagulation and platelet function and postoperative bleeding in a series of patients undergoing cardiac surgery.

Design This is a prospective cohort study. 57 adult patients presented for elective cardiac surgery were recruited in the study. Informed consent was obtained by all patients. Exclusion criteria were defined as follows: unwillingness to participate, preoperative platelet count ⩽150 × 109/mm3, age <18 or >79 years, emergency procedure, redo surgery, a known coagulation disorder and inaccurate documentation of preoperative antiplatelet medication.

Methods All patients were managed by the same surgical team and anaesthesiologist. They all received general anaesthesia in accordance with our institutional protocol. A dose of 15mg/kg tranexamic acid was given at induction of anaesthesia and after protamine administration. Surgery was performed under normothermia using a standard median sternotomy and MiECC modular (Type IV) circuit was used in all patients during CPB. An activated clotting time (ACT) value >300sec was aimed for patients undergoing CABG and an ACT>400sec for all other valve or complex surgery. Reversal of heparin was accomplished with protamine at a heparin-protamine titration ratio of 0.75.

Preoperatively demographics, comorbidities, use of anticoagulants, antiplatelet medication were collected and intraoperatively type of operation, duration of CPB, duration of aortic cross-clamp, and heparin and protamine doses were recorded. Fibrinogen levels (mg/dL) were measured before surgery (baseline) and after arrival in the ICU. Postoperative bleeding at 12 and 24 hours, as defined according to the universal definition of bleeding, was recorded, as well as intraoperative and 24-hour transfusion requirements (including blood products or coagulation factors concentrates) and major adverse events.

Platelet aggregation was measured on two time points: T1 = arriving in operating room before any drug or fluid administration and T2' = 20 minutes after heparin reversal with protamine, in whole hirudin containing blood samples using the ROTEM platelet (TEM International GmbH, Munich, Germany), which evaluates impedance aggregometry. Specific reagents were chosen: 1. adenosine diphosphate (ADP) known as ADPtest to evaluate ADP function and thienopyridine efficiency, 2. thrombin receptor activating peptide (TRAP) known as TRAPtest assay for assessment of blockage of GPIIb/IIIa or protease-activated receptor (PAR). Abnormal values were indicative of platelet dysfunction. Regarding thromboelastometry, parameters that were recorded included the EXTEM and the FIBTEM assay. EXTEM and FIBTEM assays were performed at two time points: T1: before anaesthesia induction and fluid administration and T2: after removal of aortic cross clamp. Clotting time (CT) reflecting initiation of the clotting cascade and clot formation time (CFT) reflecting fibrin polymerization and clot stabilization were measured in EXTEM assay. Maximum clot firmness (MCF), indicating clot strength, was measured in EXTEM and FIBTEM assays.

Statistical Analysis Plan The SPSS v.25.0 software (SPSS, Inc., Chicago, Ill, USA) was utilized for all statistical analyses. The significance level was set at p≤0.05 for the tested hypotheses. Continuous variables are presented as mean and standard deviation (SD). Categorical variables are expressed as absolute values and relative frequencies. Measures at the two time points were assessed for normality using the Kolmogorov Smirnov and Shapiro-Wilk tests and then analyzed with paired samples t-test or Wilcoxon U-test, as appropriate. For continuous variables, correlations were examined with Pearson or Spearman correlation according to the distribution of the data. Regression was performed for the primary outcome variables. A binary logistic regression model was used to estimate the multivariate predictive ability of perioperative variables on the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery

Exclusion Criteria:

* unwillingness to participate
* preoperative platelet count ≤150 × 109/mm3
* redo surgery
* a known coagulation disorder
* inaccurate documentation of preoperative anti-platelet medication.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at AHEPA University Hospital for cardiac surgery
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change of Clotting Time | Sample 1: baseline, Sample 2: after aortic cross clamp off
  A parameter of the EXTEM and FIBTEM test performed using Rotational Thromboelastometry (ROTEM delta,Tem Systems Inc., Munich, Germany). It is measured in seconds and was tested in two time points. Sample 1: baseline, upon admission in the operation room and Sample 2: after aortic cross clamp off.
Change of Maximum Clot Firmness | Sample 1: baseline, Sample 2: after aortic cross clamp off
  A parameter of the EXTEM and FIBTEM test performed using Rotational Thromboelastometry (ROTEM delta,Tem Systems Inc., Munich, Germany). It is measured in millimeters and was tested in two time points. Sample 1: baseline, upon admission in the operation room and Sample 2: after aortic cross clamp off.
Change of Clot Formation Time | Sample 1: baseline, Sample 2: after aortic cross clamp off
  A parameter of the EXTEM and FIBTEM test performed using Rotational Thromboelastometry (ROTEM delta,Tem Systems Inc., Munich, Germany). It is measured in seconds and was tested in two time points. Sample 1: baseline, upon admission in the operation room and Sample 2: after aortic cross clamp off.
Change of ADPtest of Impedance Aggregometry | Sample 1: baseline, Sample 2': 20 minutes after heparin reversal
  ADPtest was performed using impedance aggregometry. Results expressed with the area under the curve (AUC) and represent the area under the aggregation curve, from the start of the measurement until 6 minutes (test duration). AUC was recorded as Ohm × minutes for each test. Both tests were performed at two time points. Sample 1: baseline, upon admission in the operation room and Sample 2: 20 minutes after heparin reversal.
Change of TRAPtest of Impedance Aggregometry | Sample 1: baseline, Sample 2': 20 minutes after heparin reversal
  TRAPtest was performed using impedance aggregometry. Results expressed with the area under the curve (AUC) and represent the area under the aggregation curve, from the start of the measurement until 6 minutes (test duration). AUC was recorded as Ohm × minutes for each test. Both tests were performed at two time points. Sample 1: baseline, upon admission in the operation room and Sample 2: 20 minutes after heparin reversal.

SECONDARY OUTCOMES:
Bleeding in the drainage at 12 hours postoperatively | 12 hours after the end of the procedure
  Cumulative bleeding in the drainage
Bleeding in the drainage at 24 hours postoperatively | 24 hours after the end of the procedure
  Cumulative bleeding in the drainage
Transfusion requirements | perioperatively and during first 24h in ICU
  The transfusion requirements during surgery and during the first 24 hours in the Intensive Care Unit of each of the following were recorded:
  * Red Blood Cell Units (measured in Units),
  * Fresh Frozen Plasma Units (measured in Units),
  * Platelets Units (measured in Units).
Transfusion requirements | perioperatively and during first 24h in ICU
  The transfusion requirements during surgery and during the first 24 hours in the Intensive Care of Prothrombin Complex Concentrate (measured in International Units).
Transfusion requirements | perioperatively and during first 24h in ICU
  The transfusion requirements during surgery and during the first 24 hours in the Intensive Care of Fibrinogen Concentrate (measured in grams).
Mortality | 30 days
  death
Morbidity | 30 days
  Tracheostomy, Ischemic Cerebral Disease

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Anastasiadis, Prof, Study Chair — Director of Cardiothoracic Department, AHEPA University Hospital
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No